CLINICAL TRIAL: NCT06648733
Title: Improving Pharmacological Transition of Palliative Care Patients From Inpatient to Outpatient Care (Optimierung Der Pharmakologischen Überleitung Von Palliativpatient:Innen Von stationär Nach Ambulant)
Brief Title: Improving Pharmacological Transition of Palliative Care Patients From Inpatient to Outpatient Care
Acronym: EntMedPall
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: University Hospital Munich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-258-f-S; 2025-131-BO (Other: Ethikkommission an der Medizinischen Fakultät Bonn)
Record Dates: First submitted 2024-06-27; First posted 2024-10-18 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Heart Failure; COPD
Keywords: Palliative Care
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective patients (Experimental): Current palliative care patients who are discharged from the University Hospital to outpatient palliative care.
  Interventions: Other: Structured pharmaceutical discharge management
- Retrospective patients (No Intervention): Former palliative care patients who were discharged from the university hospital to outpatient palliative care.

INTERVENTIONS:
Other: Structured pharmaceutical discharge management — These patients will receive structured pharmaceutical discharge management from inpatient to outpatient care.
  Arms: Prospective patients

SUMMARY:
The transition of palliative care patients from inpatient to outpatient care is aimed to be improved through structured pharmaceutical discharge management by a trained pharmacist. This data will be compared with retrospective cases.

DETAILED DESCRIPTION:
As part of a prospective observational study with a retrospective comparison group, a pharmacist should, on request, check the discharge medication planned by the primary care physicians before discharge and discuss it with the various colleagues providing (follow-up) care. In addition, the availability in the outpatient "medicine cabinet" and the possibility of prescribing by the responsible GPs (by telephone) should be checked in advance. In addition, longitudinal focus groups with relevant stakeholders are to be conducted to collect quantitative data as well as qualitative data on the views of those providing and receiving treatment.

There will be cooperation with the Specialized Outpatient Palliative Care Service Muenster to ensure sufficient case numbers and a low rate of missing values through partial use of the standard care data from the "Information System Palliative Care" (ISPC) program they use.

ELIGIBILITY:
Inclusion Criteria:

All individual indications for general and specialised palliative care as part of routine clinical practice (e.g.):

* advanced, malignant tumour disease
* advanced, chronic obstructive pulmonary disease
* Patients with advanced disease and limited life expectancy (approx. 12 months) Further care in the SOPC Muenster (prospective data) Sufficient understanding of the German language to be able to understand the information and consent form

Exclusion Criteria:

Impossibility of understanding the information and declaration of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
(I) Drug-related problems | 12 months
  (I) Number of drug-related problems at the time of discharge according to PCNE (comparison of prospective, actually proposed changes vs. hypothetical number and type of problems at the time of discharge in the retrospective comparison cohort)
(II) Drug-related problems | 12 months
  (II) Type of drug-related problems at the time of discharge according to PCNE (comparison of prospective, actually proposed changes vs. hypothetical number and type of problems at the time of discharge in the retrospective comparison cohort)

SECONDARY OUTCOMES:
Number of contacts | 12 months
  Number of contacts made by patients/relatives with SOPC within 7 days of discharge
Number of readmissions / visits | 12 months
  Number of readmissions and / or visits to the emergency department within 7 and 14 days after hospital discharge
Symptom burden | 12 months
  Change in patient symptom burden via Integrated Palliative Care Outcome. The total scores using the IPOS can range between 0 and 68 points. The higher the score, the more severe are the patient's symptoms. Scale after 3, 7 and 14 days compared to day 0 (discharge date)
(I) Medication changes | 12 months
  (I) Number of medication changes suggested by pharmacists according to PCNE
Adoption rate | 12 months
  Adoption rate by the primary care physicians of the pharmacist's proposed changes after PCNE (see primary endpoint)
(I) GP contact | 12 months
  (I) Contact made with GPs for medication planning
(I) SOPC contact | 12 months
  (I) Contact made with SOPC for medication planning and (II) resulting changes to discharge medication
(I) Post-discharge medication changes | 12 months
  Change in the number of medications in outpatient follow-up care
Focus groups | 12 months
  Satisfaction of inpatient physicians and those providing further treatment with forward-looking medication planning in 3 focus groups
(I) Further parameters | 12 months
  (I)Evaluation of further quantitative parameters from ISPC (SOPC)
(II) Medication changes | 12 months
  (II) Type of medication changes suggested by pharmacists according to PCNE
(II) GP contact | 12 months
  (II) Resulting changes to discharge medication following GP contact
(II) SOPC contact | 12 months
  (II) Resulting changes to discharge medication following SOPC contact
(II) Post-discharge medication changes | 12 months
  (II) Qualitative assessment of medication changes (classification of drug-related problems according to PCNE)
(II) Further parameters | 12 months
  (II) Evaluation of further quantitative parameters from the clinical information system (UKM)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Klaas, Dr. rer. nat., Study Chair — Pharmacy of the University Hospital Muenster
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany